CLINICAL TRIAL: NCT01033370
Title: A Safety and Efficacy Study of Blood Pressure Control in Acute Aortic Emergencies - A Pilot Study (PROMPT)
Acronym: PROMPT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Project lacked funding.
Sponsor: Asma Zainab, M.D. (Other)
Collaborators: The Medicines Company (Industry); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Asma Zainab, M.D., Sponsor-Investigator/Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00003478; IRB(2)0809-0120 (Other: HMRI IRB)
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Aortic Aneurysm; Aortic Disease
Keywords: acute; aortic; emergencies; Aortic dissection
MeSH Terms: conditions — Aortic Aneurysm; Aortic Diseases; Emergencies; Aortic Dissection | interventions — clevidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label, non-randomized, pilot study (Other): All subjects who provide consent for trial participation with an acute aortic emergency and elevated BP (systolic blood pressure [SBP] ≥120 mm Hg) requiring IV antihypertensive therapy for up to 48 hours will be administered an infusion of clevidipine to evaluate the efficacy and safety of the IV drug.
  Interventions: Drug: clevidipine.

INTERVENTIONS:
Drug: clevidipine. — Clevidipine administered per IV infusion, starting dose of 2 mg/h (4 mL/hr) for 3 minutes & titrated to the desired BP lowering effect to SBP goal of < 120 mmHg, max infusion rate may not exceed 32 mg/h (64 mL/hr).
  Other Names: CLEVIPREX® (clevidipine)

SUMMARY:
This study is a single center, non-randomized, open-label, pilot efficacy and safety study evaluating the ability of clevidipine IV antihypertensive to rapidly control elevated blood pressure (BP) in the setting of an acute aortic emergencies (aneurysm, dissection or other aortic disease).

DETAILED DESCRIPTION:
This study will be a Phase IV, open label, non-randomized efficacy and safety pilot trial in patients with AAE and hypertension requiring parenteral antihypertensive therapy. For the purpose of this study hypertension is defined as SBP ≥120 mm Hg immediately prior to clevidipine administration.

Patients will be enrolled at the Methodist DeBakey Heart & Vascular Center in Houston, TX. Enrollment of approximately 30 patients is anticipated and enrollment will continue until this goal is met.

The study will include three separate periods: Screening Period, Treatment Period (up to 48 hours) and Follow-up Period (up to 7 days or hospital discharge, whichever occurs first) representing approximately a maximum of 7 days on study. Eligible patients will be enrolled to receive clevidipine IV antihypertensive treatment (study drug) in an open label manner.

Clevidipine will be infused at an initial rate of 2 mg/h (4 mL/hr) for the first 3 minutes. Thereafter, titration to higher infusion rates can be attempted as needed to obtain the target SBP goal < 120 mmHg. Titration to effect is to proceed by doubling the dose every 3 minutes, up to a maximum of 32 mg/h (64 mL/hr), until the SBP < 120 mmHg is attained.

If the desired BP lowering effect is not attained with study drug within 1 hour or not maintained thereafter, an alternative antihypertensive agent may be used, with or without stopping clevidipine IV antihypertensive infusion. The alternative agent should be used per institutional treatment practice. During the initial 1 hour of the treatment period, however, clevidipine IV antihypertensive treatment should be administered as monotherapy until 1 hour post initiation of study drug. The use of an alternative antihypertensive agent(s) is discouraged and limited to where medically necessary to maintain patient safety.

Clevidipine IV antihypertensive infusion may continue for a maximum of 48 hours. However, if medically warranted, clevidipine treatment may continue beyond 48 hours at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of AAE (aneurysm, dissection or other aortic disease)
* Baseline SBP (immediately prior to initiation of study drug) of ≥120 mm Hg
* Requires IV antihypertensive therapy to lower BP
* Written informed consent before initiation of any study related procedures

Exclusion Criteria:

* Intolerance or allergy to calcium channel blockers, soy or egg products
* Chest pain and/or electrocardiogram (ECG) with ST segment changes consistent with cardiac ischemia
* Cardiogenic shock
* Severe arrhythmia
* Severe aortic stenosis
* Positive pregnancy test, known pregnancy or breast feeding female
* Known liver failure, cirrhosis or pancreatitis
* Prior directives against advanced life support (no code status)
* Those, in the opinion of the participating physician, regarding as inappropriate for the study for any other medical reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of this pilot study is to evaluate the efficacy of an IV infusion of clevidipine as an antihypertensive for BP lowering in patients with AAE and elevated BP. | 1 Hour

SECONDARY OUTCOMES:
The secondary objectives of the study are to evaluate the safety of an IV infusion of clevidipine as an antihypertensive for BP lowering in patients with AAE and elevated BP. | 48 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Masud, MD, Principal Investigator — The Methodist Hospital and The Methodist Hospital Research Institute; Asma Zainab, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- The Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Incomplete data set due to early trial closure.

REFERENCES:
- [Background] Clevidipine Investigator's Brochure, 2009.
- [Background] Cleviprex Prescribing Information, August 1, 2008
- [Background] Cheung AT, Hobson RW 2nd. Hypertension in vascular surgery: aortic dissection and carotid revascularization. Ann Emerg Med. 2008 Mar;51(3 Suppl):S28-33. doi: 10.1016/j.annemergmed.2007.11.011. Epub 2008 Jan 11. No abstract available. PMID 18191301
- [Background] Kertai MD, Westerhout CM, Varga KS, Acsady G, Gal J. Dihydropiridine calcium-channel blockers and perioperative mortality in aortic aneurysm surgery. Br J Anaesth. 2008 Oct;101(4):458-65. doi: 10.1093/bja/aen173. Epub 2008 Jun 12. PMID 18556693
- [Background] Golledge J, Eagle KA. Acute aortic dissection. Lancet. 2008 Jul 5;372(9632):55-66. doi: 10.1016/S0140-6736(08)60994-0. PMID 18603160
- [Background] Khoynezhad A, Plestis KA. Managing emergency hypertension in aortic dissection and aortic aneurysm surgery. J Card Surg. 2006 Mar-Apr;21 Suppl 1:S3-7. doi: 10.1111/j.1540-8191.2006.00213.x. PMID 16492293
- [Background] Suzuki T, Mehta RH, Ince H, Nagai R, Sakomura Y, Weber F, Sumiyoshi T, Bossone E, Trimarchi S, Cooper JV, Smith DE, Isselbacher EM, Eagle KA, Nienaber CA; International Registry of Aortic Dissection. Clinical profiles and outcomes of acute type B aortic dissection in the current era: lessons from the International Registry of Aortic Dissection (IRAD). Circulation. 2003 Sep 9;108 Suppl 1:II312-7. doi: 10.1161/01.cir.0000087386.07204.09. PMID 12970252
- [Background] Mehta RH, Suzuki T, Hagan PG, Bossone E, Gilon D, Llovet A, Maroto LC, Cooper JV, Smith DE, Armstrong WF, Nienaber CA, Eagle KA; International Registry of Acute Aortic Dissection (IRAD) Investigators. Predicting death in patients with acute type a aortic dissection. Circulation. 2002 Jan 15;105(2):200-6. doi: 10.1161/hc0202.102246. PMID 11790701
- [Background] Erbel R, Alfonso F, Boileau C, Dirsch O, Eber B, Haverich A, Rakowski H, Struyven J, Radegran K, Sechtem U, Taylor J, Zollikofer C, Klein WW, Mulder B, Providencia LA; Task Force on Aortic Dissection, European Society of Cardiology. Diagnosis and management of aortic dissection. Eur Heart J. 2001 Sep;22(18):1642-81. doi: 10.1053/euhj.2001.2782. No abstract available. PMID 11511117
- [Background] Hagan PG, Nienaber CA, Isselbacher EM, Bruckman D, Karavite DJ, Russman PL, Evangelista A, Fattori R, Suzuki T, Oh JK, Moore AG, Malouf JF, Pape LA, Gaca C, Sechtem U, Lenferink S, Deutsch HJ, Diedrichs H, Marcos y Robles J, Llovet A, Gilon D, Das SK, Armstrong WF, Deeb GM, Eagle KA. The International Registry of Acute Aortic Dissection (IRAD): new insights into an old disease. JAMA. 2000 Feb 16;283(7):897-903. doi: 10.1001/jama.283.7.897. PMID 10685714